CLINICAL TRIAL: NCT02710591
Title: A Phase Ib, Open Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Oral Doses of Rimeporide in Patients With Duchenne Muscular Dystrophy
Brief Title: Rimeporide in Patients With Duchenne Muscular Dystrophy
Acronym: RIM4DMD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EspeRare Foundation (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EspeRare_RIM_001; 2015-002530-50 (EudraCT Number)
Record Dates: First submitted 2016-01-26; First posted 2016-03-17 (Estimated); Results first posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-01

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Rimeporide
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — N-(2-methyl-4,5-bis(methylsulfonyl)benzoyl)guanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rimeporide (Experimental): Multiple oral doses of rimeporide ranging from 50 to 300 mg will be administered three times a day (TID) for a total of 4 weeks. 4 ascending dose levels will be studied sequentially in ascending order. Rimeporide is provided as hard gel 25 mg or 50 mg capsules.
  Each patient will participate in only 1 dose cohort. 5 patients are expected to be recruited in each cohort through all participating sites.
  Interventions: Drug: Rimeporide

INTERVENTIONS:
Drug: Rimeporide — Cohort 1:
  50 mg TID in patients with a body weight ≤ 30kg at Baseline and 75 mg TID in patients with a body weight > 30kg at Baseline
  Cohort 2:
  100mg TID in patients with a body weight ≤ 30kg at baseline and 150 mg TID in patients with a body weight > 30kg at Baseline
  Cohort 3:
  150 mg TID in patients with a body weight ≤ 30kg at baseline and 200 mg TID in patients with a body weight > 30kg at Baseline
  Cohort 4:
  200 mg TID in patients with a body weight ≤ 30kg at Baseline and 300 mg TID mg TID in patients with a body weight > 30kg at Baseline
  Other Names: EMD 87580

SUMMARY:
In Duchenne Muscular Dystrophy (DMD) there is an imbalance between the levels of calcium and sodium in the muscles cells which is thought to be important in the damage which occurs overtime. Sodium/proton type 1 exchanger (NHE-1) inhibition is an innovative pathway that has proved to efficiently prevent the accumulation of muscle damage (inflammation and fibrosis) in animal models of muscular dystrophies and heart failure. Based on prior safety and efficacy results in animal and humans, NHE-1 inhibition with Rimeporide represents a new therapeutic approach with no restriction on age and on genetic subtypes which could be combined to other treatments that restore or augment dystrophin.This study examines the safety and tolerability and effects on the muscles of rimeporide, in patients aged 6 to 14 years with Duchenne Muscular Dystrophy (DMD).

DETAILED DESCRIPTION:
This study is designed as a phase Ib, multicenter, european, open label study to evaluate the safety and tolerability and biomarkers of a new drug, rimeporide, in boys aged 6 to 14 years with Duchenne Muscular Dystrophy (DMD).

Rimeporide will be taken orally for 4 weeks, three times a day. Dose will be adapted to body weight. The study will enrol 20 patients with DMD, aged 6 to 14 years. 4 dose levels will be tested, in 4 different cohorts with 5 patients taking the drug at each dose level.

During the study, there will be 6 visits in the Hospital over a maximum of 10 weeks. At each visit, patients will undergo safety examinations including vital signs, physical and neurological examinations, ECG, safety and hematology, biochemistry and urinalysis, concomitant treatments review, and any symptoms and side effects review. In addition, blood samples will be withdrawn for the evaluation of Rimeporide in plasma. Finally, additional blood & urine samples will be collected to explore efficacy markers. Patients will also undergo 2 NMR (at screening and End of study) to develop non invasive biomarkers for further investigations in DMD patients.

The decision to progress to the next higher dose will be made after safety and tolerability data are reviewed for the preceding dose for 5 patients by SMC and determined that it is safe to proceed to the next dose level.

ELIGIBILITY:
Inclusion Criteria:

* Duchenne muscular dystrophy genetically confirmed;
* Males between 6 and 14 years old;
* Able to walk independently at least 75 meters;
* Patients on a stable dose of corticosteroids at least 6 months prior to baseline;
* Patients able to swallow capsules size 4 according to the parents and investigator opinion;
* Willing and able to comply with all protocol requirements and procedures;
* Signed informed consents by the parent(s)/legal guardian(s);
* France only: Affiliated to or a beneficiary of a social security system

Exclusion Criteria:

* Patients with significant renal disease or impairment, with Glomerular Filtration Rate estimated using plasma cystatin C level using the Filler formula less than 90ml/min/1.73m2
* Current or history of liver disease or impairment,
* History of any significant medical disorder which may confound the interpretation of either efficacy or safety data e.g. inflammatory, coagulation disease, unstable cardiac or respiratory disease
* Acute illness within 4 weeks of the first administration of study medication which may interfere with study assessments;
* Significant change of dosage and/or dosing regimens for corticosteroids planned for the duration of study medication;
* Use of beta blockers / and ACEI or ARB unless at stable dose for at least 3 months prior to baseline;
* Use of Proton Pump Inhibitors unless at a stable dose for at least 3 months prior to baseline
* Use of aldosterone antagonists (i.e. spironolactone, eplerenone) within 3 months prior to first administration of study medication;
* Use of anticoagulants, antithrombotics or antiplatelet agents,
* Use of antibiotics with predominant renal secretion (e.g., cephalosporins), immunosuppressive agents exception corticosteroids, continuous treatment with non-steroidal, anti-inflammatory drugs (NSAIDs), or lithium;
* Previous treatment with idebenone or other forms of Coenzyme Q10 within 1 month of the first administration of study medication;
* Previous treatment with investigational drugs within 4 weeks (or 7 half-life if longer than 4 weeks) of the first administration of study medication including placebo;
* A baseline QTc>450msec,or history of risk factors for torsades de pointes (eg, heart failure, hypokalaemia, family history of long QT syndrome);
* LVEF≤ 45% at screening or within the past 6 months and/or history of acute heart failure;
* Ventilator dependent;
* Known individual hypersensitivity to any of the ingredients/excipients of the study medication;
* Patients with specific contraindication to MRI (e.g.: metallic foreign body, claustrophobia, etc.).

Ages: 6 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Porte-Thomé, Study Director — R&D Director EspeRare
Locations (4):
- I-Motion - Hôpital Armand Trousseau, Paris, Île-de-France Region, France
- San Raffaele Hospital, Milan, Italy
- Santa Creu i Sant Pau Hospital, Barcelona, Spain
- UCL Institute of Child Health and Great Ormond Street Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — http://esperare.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period varied depending on the recruitment speed ; started in March 2016 to November 2017. it was competitive among the 4 sites: France, Spain, Italy and UK. A time interval of at least 1 week was maintained between adminstration of first dose in the first 3 patients of each cohort. It was extended to all patients for cohort 4.
Pre-assignment Details: Screening details:
  Screening was carried out within 4 week prior to first administration of Rimeporide (SD1) to enable confirmation of patient eligibility and following the signature of the Informed Consent Form.
Groups:
- Cohort 1: 5 patients in total: patients with a body weight less than or equal to 30kg at baseline were administered 50 mg TID; patients with a body weight more than 30kg at baseline were administered 75 mg TID. Each patient received Rimeporide during 4 weeks.
- Cohort 2: 5 patients in total: patients with a body weight less than or equal to 30kg at baseline were administered 100 mg TID; patients with a body weight more than 30kg at baseline were administered 150 mg TID. Each patient received Rimeporide during 4 weeks.
- Cohort 3: 5 patients in total: patients with a with a body weight less than or equal to 30kg at baseline were administered 150 mg TID; patients with a body weight more than 30kg at baseline were administered 200 mg TID. Each patient received rimeporide during 4 weeks.
- Cohort 4: 5 patients in total: patients with a body weight less than or equal to 30kg at baseline were administered 200 mg TID; patients with a body weight more than 30kg at baseline were administered 300 mg TID. Each patient received rimeporide during 4 weeks
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population (all patients receiving at least one dose of Rimeporide)
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 5 | 5 | 5 | 20
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (1.7) | 8.2 (1.5) | 8.8 (1.6) | 9.2 (0.4) | 8.7 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 5 | 5 | 5 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 5 | 5 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 0 | 1 | 3 | 1 | 5
  Italy | 0 | 1 | 2 | 3 | 6
  France | 5 | 0 | 0 | 1 | 6
  Spain | 0 | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Observations are given for the safety population (all patients who received at least one dose of study drug). Categorical data are presented with the number of subjects with at least one event for the following selections:
  * treatment-emergent AEs (TEAEs)
  * study drug-related TEAEs (ADRs)
  * serious TEAEs
  * study drug-related serious TEAEs (serious ADRs)
  * TEAEs leading to withdrawal
  * study drug-related TEAEs (ADRs) leading to withdrawal
  * serious TEAEs leading to withdrawal
  * TEAEs leading to death as outcome
Time Frame: up to 6 weeks from first administration
Population: Observations are given for the safety population (all patients who received at least one dose of study drug).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 5 | 5 | 5
Participants
  Treatment emergent adverse events (TEAEs) | 2 | 1 | 5 | 4
  Treatment emergent adverse drug reactions (ADRs) | 0 | 0 | 0 | 2
  SAEs | 0 | 0 | 1 | 0
  Serious ADRs | 0 | 0 | 0 | 0
  TEAEs leading to withdrawal | 0 | 0 | 0 | 0
  TEAEs leading to death | 0 | 0 | 0 | 0

2. Other Pre Specified Outcome: PK Profile of Rimeporide - Cmax
Description: PK samples were collected according to the following schedule:
  * At Day 1: for half of the patients: just before first administration, and one sample in each of the following time frames after the first dose:
    * 0.5 to 1h after dosing,
    * 1 to 2h after dosing,
    * 2.5 to 3.5h after dosing,
    * 6h after dosing
  * At Day 1: for the other half of the patients: just before first administration, and one sample in each of the following time frames after the second dose:
    * 0.5 to 1h after dosing,
    * 1 to 2h after dosing,
    * 2.5 to 3.5h after dosing,
    * 6h after dosing
  Finally, at week 4 (Day 28) after the last dose:
  * 0.5 to 1h after dosing,
  * 6h after dosing
Time Frame: 4 week study treatment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 5 | 5 | 5 | 5
ng/mL
  Cmax at Day 1 | 1286 (568) | 1987 (650) | 3013 (730) | 3819 (743)
  Cmax at Day 28 | 1361 (431) | 2077 (974) | 2817 (675) | 3909 (846)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from first administration of the study drug up to 6 weeks.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 1/5 | 5/5 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=5) | Cohort 3 (N=5) | Cohort 4 (N=5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=5) | Cohort 2 (N=5) | Cohort 3 (N=5) | Cohort 4 (N=5)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT02710591/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT02710591/SAP_001.pdf